CLINICAL TRIAL: NCT06344104
Title: A Double-Blind, Randomised, Placebo-Controlled, Multicentre Study Evaluating the Efficacy and Safety of Baxdrostat in Participants With Uncontrolled Hypertension on Two or More Medications Including Participants With Resistant Hypertension
Brief Title: A Study to Investigate the Efficacy and Safety of Baxdrostat in Participants With Uncontrolled Hypertension on Two or More Medications Including Participants With Resistant Hypertension
Acronym: BaxAsia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6970C00008
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Uncontrolled Hypertension; Resistant Hypertension
Keywords: Hypertension; Uncontrolled hypertension; Resistant hypertension; Blood pressure; Baxdrostat; CIN-107; Aldosterone; Aldosterone synthase
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 mg baxdrostat (Experimental): 2 mg baxdrostat administered orally, once daily (QD)
  Interventions: Drug: Baxdrostat
- 1 mg baxdrostat (Experimental): 1 mg baxdrostat administered orally, once daily (QD).
  Interventions: Drug: Baxdrostat
- placebo (Placebo Comparator): Placebo administered orally, once daily (QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat tablet administered orally, once daily (QD). Unit dose strength:
  * 1 mg per tablet for 1mg baxdrostat Arm
  * 2 mg per tablet for 2mg baxdrostat Arm
  Other Names: CIN-107
  Arms: 1 mg baxdrostat; 2 mg baxdrostat
Drug: Placebo — Placebo tablet administered orally, once daily (QD).
  Arms: placebo

SUMMARY:
The purpose of this study is to measure the efficacy and safety of baxdrostat in participants with uHTN or rHTN. The main objective is to compare the difference in SBP change from baseline at Week 12 of treatment between participants receiving 2 mg baxdrostat or 1 mg baxdrostat tablets and participants receiving placebo tablets.

DETAILED DESCRIPTION:
This is a Phase III, multicentre, randomised, double-blinded, placebo-controlled, parallel group study to evaluate the safety, tolerability and effect of 1 or 2 mg baxdrostat versus placebo, administered QD orally, on the reduction of SBP in approximately 300 participants aged ≥ 18 years with HTN (≥ 140 mmHg at Screening; ≥ 135 mmHg at randomisation) despite a stable regimen of 2 antihypertensive agents at baseline, one of which is a diuretic (uHTN); or ≥ 3 antihypertensive agents at baseline, one of which is a diuretic (rHTN).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be ≥ 18 years old.
* Mean seated SBP on automated office blood pressure measurement (AOBPM) ≥ 140 mmHg at Screening.
* Fulfil at least 1 of the following 2 criteria:

  1. uHTN subpopulation: have a stable regimen (≥ 4 weeks) of 2 antihypertensive medications, from different therapeutic classes (at least one must be a diuretic), at maximum tolerated dose in the judgement of the Investigator.
  2. rHTN subpopulation: have a stable regimen (≥ 4 weeks) of ≥ 3 antihypertensive medications, from different therapeutic classes (at least one must be a diuretic), at maximum tolerated dose in the judgement of the Investigator.
* Estimated glomerular filtration rate ≥ 45 mL/min/1.73m2 at Screening.
* Serum potassium (K+) level ≥ 3.5 and < 5.0 mmol/L at Screening.• Mean seated SBP on AOBPM ≥ 135 mmHg at Baseline.

Exclusion Criteria:

* Mean seated SBP on AOBPM ≥ 170 mmHg.
* Mean seated DBP on AOBPM ≥ 105 mmHg.
* Serum sodium level (Na+) < 135 mmol/L at Screening.
* Has the following known secondary causes of hypertension: renal artery stenosis, uncontrolled or untreated hyperthyroidism, uncontrolled or untreated hypothyroidism, pheochromocytoma, Cushing's syndrome, aortic coarctation.
* NYHA functional heart failure class IV at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in seated SBP at Week 12 | At Week 12
  To assess the effect of 2 mg baxdrostat versus placebo on seated SBP at Week 12

SECONDARY OUTCOMES:
Change from baseline in seated SBP at Week 12 | At Week 12
  To assess the effect of 1 mg baxdrostat versus placebo on seated SBP at Week 12
Change from RWD baseline (Week 24) in seated SBP at Week 32 | At Week 32
  To assess the effect of 2 mg baxdrostat versus placebo on seated SBP at 8 weeks after randomised withdrawal
Change from baseline in the mean ambulatory 24-hour SBP at Week 12 as measured by ABPM | At Week 12
  To assess the effect of treatment with baxdrostat 2 mg vs placebo on ambulatory 24-hour average SBP at Week 12
Change from baseline in the mean ambulatory 24-hour SBP at Week 12 as measured by ABPM | At Week 12
  To assess the effect of treatment with baxdrostat 1 mg vs placebo on ambulatory 24-hour average SBP at Week 12
Change from baseline in seated DBP at Week 12 | At Week 12
  To assess the effect of 2 mg baxdrostat versus placebo on seated DBP at Week 12
Achieving seated SBP < 140 mmHg at Week 12 | At Week 12
  To assess the effect of 2 mg baxdrostat versus placebo on achieving seated SBP < 140 mmHg at Week 12
Change from baseline in seated DBP at Week 12 | At Week 12
  To assess the effect of 1 mg baxdrostat versus placebo on seated DBP at Week 12
Achieving seated SBP < 140 mmHg at Week 12 | At Week 12
  To assess the effect of 1 mg baxdrostat versus placebo on achieving seated SBP < 140 mmHg at Week 12
Change from baseline in seated SBP at Week 12 | At Week 12
  To assess the effect of 2 mg baxdrostat versus placebo on seated SBP at Week 12 in the rHTN subgroup
Change from baseline in seated SBP at Week 12 | At Week 12
  To assess the effect of 1 mg baxdrostat versus placebo on seated SBP at Week 12 in the rHTN subgroup

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | Up to week 54
  To assess the safety and tolerability of baxdrostat versus placebo. Occurrence of adverse events (AE), including serious adverse events (SAEs), adverse events leading to treatment discontinuation (DAE) and adverse events of special interest (AESI)

CONTACTS AND LOCATIONS:
Locations (73):
- Argentina (5):
  - Research Site, Bahía Blanca
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás de los Arroyos
- Australia (4):
  - Research Site, Coffs Harbour
  - Research Site, Gosford
  - Research Site, Hoppers Crossing
  - Research Site, Ipswich
- China (32):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Deyang
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Ha’erbin
  - Research Site, Hefei
  - Research Site, Heze
  - Research Site, Jiujiang
  - Research Site, Luoyang
  - Research Site, Meihekou
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Panjin
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xianyang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zigong
- Research Site, Hong Kong, Hong Kong
- India (2):
  - Research Site, Bangalore
  - Research Site, Belagavi
- Japan (11):
  - Research Site, Chūōku
  - Research Site, Hamamatsu
  - Research Site, Kagoshima
  - Research Site, Koga-shi
  - Research Site, Meguro-ku
  - Research Site, Minatoku
  - Research Site, Minokamo Shi
  - Research Site, Osaka
  - Research Site, Toshima-ku
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Philippines (2):
  - Research Site, Iloilo City
  - Research Site, Quezon City
- Russia (3):
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Seoul, South Korea
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Kahramanmaraş
  - Research Site, Karşıyaka
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Mersin
- Vietnam (5):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/